CLINICAL TRIAL: NCT00331305
Title: Exercise Training and Depression in Older Adults II
Brief Title: Exercise Training Versus Drug Therapy for Treating Depression in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00010275; R01MH049679 (NIH); DSIR GT-GS
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2007-12

CONDITIONS: Depression
Keywords: Exercise
MeSH Terms: conditions — Depression; Motor Activity | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Supervised Exercise
Behavioral: Home-Based Exercise
Drug: Sertraline (Zoloft)
Drug: Placebo Pill

SUMMARY:
This study will evaluate the effectiveness of both center-based and home-based exercise versus the antidepressant drug sertraline in treating depression in middle-aged and older adults.

DETAILED DESCRIPTION:
The combination of an aging population and the increased prevalence of chronic diseases among the elderly presents a major public health concern. Depression acts as both a cause and a consequence of disability, and with major depressive disorder (MDD) affecting up to 25% of women and 12% of men during their lifetimes, effective treatments for people of all ages must be made available. Although antidepressant medications are available as treatments for MDD, they sometimes either do not adequately relieve depressive symptoms, or do relieve depressive symptoms, but cause undesirable side effects. These side effects may become more common or more problematic as people age. Alternative approaches to treating depression, therefore, are necessary. Research suggests that exercise positively affects the levels of certain mood-enhancing neurotransmitters in the brain. This study will evaluate the effectiveness of both center-based and home-based exercise versus the antidepressant drug sertraline in treating depression in middle-aged and older adults.

Participants in this double-blind study will be randomly assigned to one of the following four treatments for 16 weeks: supervised aerobic exercise; home-based aerobic exercise; drug therapy; or placebo. All participants assigned to an exercise condition will report to the study site for a baseline exercise stress test. Participants assigned to supervised aerobic exercise will attend study visits 3 times per week for an exercise session. Each session will entail 10 minutes of warm-up exercises, followed by 30 to 35 minutes of continuous walking, biking, or jogging, and 10 to 15 minutes of cool-down exercises. Participants assigned to home-based aerobic exercise will attend one introductory session with an exercise physiologist, who will prescribe an exercise regimen and provide instruction on how to self-monitor pulse rate. They will also receive written information about their exercise plan, tips for maintaining progress and relapse prevention, and daily activity logs. The exercise prescription will be adjusted on a bi-weekly basis. Participants will be expected to exercise 3 times per week on their own, and will perform 10 minutes of warm-up exercises, followed by 30 to 35 minutes of continuous walking, biking, or jogging, and 10 to 15 minutes of cool-down exercises. In addition, they will mail in daily activity logs weekly for the first 6 weeks and biweekly for the remaining 10 weeks. Brief telephone contacts will be made to monitor progress, answer questions, and provide individualized feedback. Additionally, the exercise physiologist will conduct home visits at Weeks 4 and 8. Participants assigned to receive sertraline or placebo will receive their medication in pill-form at baseline and Weeks 2, 4, 8, 12, and 16 study visits. All participants will receive several phone calls to assess treatment response and suicide risk. These calls will take place weekly for the first 4 weeks and biweekly for the remainder of the study. Follow-up visits will occur at Months 6 and 12 post-treatment, and will include participating in psychological interviews and filling out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depressive disorder (MDD)
* Score of greater than 11 on the Beck Depression Inventory (BDI)

Exclusion Criteria:

* Primary psychiatric diagnosis other than major depressive disorder (e.g., bipolar disorder)
* Any of the following DSM-IV diagnoses: dementia or delirium; obsessive compulsive disorder (OCD); schizophrenia, schizoaffective, or other psychotic disorder; psychotic features, including any delusions or hallucinations during the current depressive episode; current alcohol or other substance abuse disorder; acute risk for suicide (e.g., score of greater than 2 on the suicide item on the HAM-D) or acute risk for homicide
* May require treatment with additional psychotherapeutic agents (other than chloral hydrate for sleep) during the course of the study
* Significant medical conditions that may cause an increased risk for a significant adverse experience during the course of the trial (e.g., unstable angina, myocardial infarction within 3 months of study entry, etc.)
* Unable to be randomly assigned to the study drug due to a risk for adverse cardiac events, such as prolonged QT interval, use of other medications that would be counterindicated for use with sertraline, or other conditions that may make study participation unsafe
* Unable to be randomly assigned to an exercise condition due to medical conditions such as musculoskeletal problems or abnormal cardiac response to exercise (e.g., exercise-induced ventricular tachycardia, abnormal blood pressure response, etc.)
* Currently receiving antidepressant medication or actively engaged in psychotherapy
* Currently exercising regularly

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 1999-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Measured at Week 16 and Months 6 and 12 post-treatment: Post-treatment recovery from MDD
Post-treatment depression scores on the Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Measured at Week 16 and Months 6 and 12 post-treatment: Quality of life (MOS SF 36)
Anxiety (State Trait Anxiety Inventory)
Cognitive Functioning (selected subtests from the Wechsler Memory Scale-R and WAIS-III; Digit Vigilance; Trail Making Test; Finger Tapping Test; Controlled Oral Word Association)
Cardiovascular biomarkers, including flow mediated dilation, heart rate variability, and baroreflex sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: James A. Blumenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Department of Psychiatry and Behavioral Sciences, Durham, North Carolina, United States

REFERENCES:
- [Background] Blumenthal JA, Babyak MA, Moore KA, Craighead WE, Herman S, Khatri P, Waugh R, Napolitano MA, Forman LM, Appelbaum M, Doraiswamy PM, Krishnan KR. Effects of exercise training on older patients with major depression. Arch Intern Med. 1999 Oct 25;159(19):2349-56. doi: 10.1001/archinte.159.19.2349. PMID 10547175
- [Background] Barbour KA, Blumenthal JA. Exercise training and depression in older adults. Neurobiol Aging. 2005 Dec;26 Suppl 1:119-23. doi: 10.1016/j.neurobiolaging.2005.09.007. Epub 2005 Oct 11. PMID 16223547
- [Derived] Sherwood A, Blumenthal JA, Smith PJ, Watkins LL, Hoffman BM, Hinderliter AL. Effects of Exercise and Sertraline on Measures of Coronary Heart Disease Risk in Patients With Major Depression: Results From the SMILE-II Randomized Clinical Trial. Psychosom Med. 2016 Jun;78(5):602-9. doi: 10.1097/PSY.0000000000000301. PMID 26867076
- [Derived] Hoffman BM, Babyak MA, Craighead WE, Sherwood A, Doraiswamy PM, Coons MJ, Blumenthal JA. Exercise and pharmacotherapy in patients with major depression: one-year follow-up of the SMILE study. Psychosom Med. 2011 Feb-Mar;73(2):127-33. doi: 10.1097/PSY.0b013e31820433a5. Epub 2010 Dec 10. PMID 21148807
- [Derived] Blumenthal JA, Babyak MA, Doraiswamy PM, Watkins L, Hoffman BM, Barbour KA, Herman S, Craighead WE, Brosse AL, Waugh R, Hinderliter A, Sherwood A. Exercise and pharmacotherapy in the treatment of major depressive disorder. Psychosom Med. 2007 Sep-Oct;69(7):587-96. doi: 10.1097/PSY.0b013e318148c19a. Epub 2007 Sep 10. PMID 17846259